CLINICAL TRIAL: NCT07129239
Title: High Dose (HD) Aflibercept Switch in Neovascular Age-related Macular Degeneration (nAMD): to Load or Maintain (HEIRLOOM)
Acronym: HEIRLOOM
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Clinique de Retine de l'est (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Dr. Andrei Szigiato, Principal Investigator, Clinique de Retine de l'est
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 23002
Record Dates: First submitted 2025-07-10; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Wet Age-related Macular Degeneration (wAMD)
MeSH Terms: interventions — Maintenance

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Loading interval group (No Intervention): patients who are currently being treated with EYLEA® (aflibercept 2mg) will be switched to EYLEA® HD (aflibercept 8mg) and receive injections every month for the first 3 months followed by an extension (or increase in dosing interval) of therapy based on clinical response. This is the "on label" treatment regimen approved by Health Canada.
- Maintenance interval group (Experimental): patients who are currently being treated with EYLEA® (aflibercept 2mg) will be switched to EYLEA® HD (aflibercept 8mg) and maintain the current treatment interval that they had with EYLEA® (aflibercept 2mg), followed by an extension of therapy (or increase in treatment dosing interval) based on clinical response. This is the "off-label" treatment regimen that we are testing to see if it is as effective and involves less treatment burden.
  Interventions: Other: Maintenance

INTERVENTIONS:
Other: Maintenance — Patients who are currently being treated with EYLEA® (aflibercept 2mg) will be switched to EYLEA® HD (aflibercept 8mg) and maintain the current treatment interval that they had with EYLEA® (aflibercept 2mg), followed by an extension of therapy (or increase in treatment dosing interval) based on clinical response
  Arms: Maintenance interval group

SUMMARY:
The purpose of this study is to compare two treatment frequencies using EYLEA® HD (aflibercept 8mg) in patients with wet age-related macular degeneration (wAMD) that are currently treated with EYLEA® (aflibercept 2mg).

EYLEA® HD is approved by Health Canada has been tested in large clinical trials involving thousands of patients around the world and has been shown effective in the treatment of wAMD. The treatment regimen used in these trials involved 3 initial monthly injections of EYLEA® HD followed by an extension of the treatment interval on the 4th visit. This was necessary since all patients in this study did not previously have treatment injections for wAMD.

Currently there is not enough information on the best treatment regimen to use for patients that are switched to EYLEA® HD from EYLEA®.

Health Canada currently recommends that EYLEA® HD is administered every month for the first 3 doses, followed by a treatment every 8 to 16 weeks.

A total of 180 patients >18 years of age will participate in this study, which will be conducted at the Clinique de Retine de l'Est in Montreal, Quebec, Canada.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18
* Patients with neovascular AMD
* Patients who have received aflibercept 2mg for a minimum of 3 loading injections plus 2 maintenance injections.
* Can include 1 or 2 eyes per patient if one or both meet study criteria.

Exclusion Criteria:

* Patients with other maculopathy, including but not limited to:
* Polypoidal choroidal vasculopathy
* Macular dystrophies (ie. Pattern dystrophy, central areolar etc.)
* Toxic/drug induced maculopathies
* Disciform scar
* Subfoveal atrophy
* Previous Photodynamic Therapy (PDT) or focal laser
* Is currently enrolled in another clinical study or observational study
* Active use of a different agent in the fellow eye, to avoid cross-over effects of anti Vascular Endothelial Growth Factor (VEGF) administration to the fellow eye
* If the patient is pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2025-08-20 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Central Retinal Thickness (CRT) | 6 and 12 month
  The primary endpoint will derived from Optical Coherence Tomography (OCT), in µm and measured at 12 months after switching therapies with interim analysis at 6 months (Detected on 8 line radial scans, through the fovea).

SECONDARY OUTCOMES:
Visual Acuity | 6 and 12 month
  Visual acuity measured by the Snellen method and then converted to Early Treatment Diabetic Retinopathy Study (EDTRS) letters. Change in visual acuity will be assessed at 6 and 12 months compared to baseline.
Number of injections | 6 and 12 month
  duration between last injection at 6 months and 12 months from date of the switch measured
Adverse events | 6 and 12 month
  Will be reported at 6 and 12 months from date of the switch measured by frequency of events (numerical), as well as descriptive for what type of adverse event.
Presence of Subretinal Fluid (Yes/No) | 6 months and 12 months
  This measure will be derived from Optical Coherence Tomography (OCT), and measured at 12 months after switching therapies with interim analysis at 6 months (Detected on 8 line radial scans, through the fovea).
Presence of Intraretinal Fluid (Yes/No) | 6 months and 12 months
  This measure will be derived from Optical Coherence Tomography (OCT), and measured at 12 months after switching therapies with interim analysis at 6 months (Detected on 8 line radial scans, through the fovea).
Pigment Epithelial Detachment (PED) Type | 6 months and 12 months
  Morphology and type of PED will be derived from Optical Coherence Tomography (OCT), and measured at 12 months after switching therapies with interim analysis at 6 months (Detected on 8 line radial scans, through the fovea).
Pigment Epithelial Detachment (PED) Height | 6 months and 12 months
  This outcome measure will be derived from Optical Coherence Tomography (OCT), measured in um, and measured at 12 months after switching therapies with interim analysis at 6 months (Detected on 8 line radial scans, through the fovea).

CONTACTS AND LOCATIONS:
Overall Officials: Andrei Szigiato, Docteur, Principal Investigator — Clinique de Retine de l'est
Locations (1):
- Clinique de Retine de L'Est, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No